CLINICAL TRIAL: NCT07212725
Title: Solving SCI Pain: Pain Recovery Tools for SCI. A 7-Week Mind/Body Self-Management Program Within a 10-Week Study
Brief Title: Solving SCI Pain: Pain Recovery Tools for SCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Spinal Cord Injury Ontario (Unknown); International Collaboration on Repair Discoveries (Other)
Responsible Party: Principal Investigator, Kathleen Martin Ginis, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI Pain Intervention - N of 1
Record Dates: First submitted 2025-08-19; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury; Pain Management; Self-management Behaviors
Keywords: Spinal Cord Injury; Chronic pain; pain interference; behaviour change; pain self-management; peer-led intervention; neuroscience-based education; body-based tools
MeSH Terms: conditions — Spinal Cord Injuries; Agnosia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: N of 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Pilot Group for Solving SCI Pain (Experimental): Participants receive a 7-week, peer-led, neuroscience-informed pain self-management program designed for individuals with SCI and chronic pain. The program includes three 2-hour virtual group education sessions covering pain neuroscience, fear-avoidance, and optional body-based tools (e.g., movement, red light therapy, percussion massage, Graston technique). Four individualized coaching sessions (up to 1 hour each) provide tailored support. Participants engage with recommended tools between sessions and complete structured check-ins every five days. Mechanism assessments (e.g., pain beliefs, self-efficacy, emotional reactivity) are conducted during the program, with full outcome measures collected at baseline, post-intervention, and follow-up. The intervention emphasizes autonomy, personal relevance, and peer support, distinguishing it from standard clinician-led approaches.
  Interventions: Behavioral: Solving SCI Pain: Peer-Led Pain Self-Management Pain Tools Program

INTERVENTIONS:
Behavioral: Solving SCI Pain: Peer-Led Pain Self-Management Pain Tools Program — Solving SCI Pain Tools is a 7-week, peer-led, neuroscience-informed pain self-management program uniquely designed for individuals with spinal cord injury (SCI) and chronic pain. It integrates cognitive and body-based tools not commonly combined in other interventions, such as red light therapy, percussion massage, Graston technique, and guided movement, alongside education on pain neurobiology and behavior change. The program is delivered virtually and emphasizes participant autonomy, optionality, and personal relevance. Distinctively, it includes multiple individualized coaching sessions led by a peer with lived experience of SCI and pain. The program does not prescribe a fixed protocol but encourages flexible, self-paced exploration supported by structured check-ins. The integration of optional, non-clinical somatic tools with behavior-change coaching and SCI-specific education distinguishes this intervention from traditional rehabilitation or pain management programs.

SUMMARY:
Brief Summary The goal of this clinical trial is to evaluate whether a neuroscience-informed, peer-led self-management program can promote behavior change and reduce pain interference in adults with spinal cord injury (SCI) and chronic pain. The primary aim is to support participants in developing practical, sustainable strategies for managing chronic pain through education, reflection, and consistent application of self-management tools. The program is designed to shift participants from passive recipients of care to active agents in their own pain management process.

Chronic pain is highly prevalent among individuals with SCI, and many report that traditional treatments - primarily pharmacological - provide limited relief and are accompanied by significant side effects. There is a growing need for accessible, non-clinical interventions that empower individuals to manage pain based on the latest neuroscience and behavior change principles.

Solving SCI Pain intervention is a 7-week, multi-component program grounded in brain-based pain science, neuroplasticity, and behavior change models. The main questions it aims to answer are:

* Does the intervention lead to meaningful changes in behavior that support pain self-management?
* Does it reduce pain interference in everyday life?

Participants will:

* Attend three 2-hour group education sessions focused on the neuroscience of pain, the role of fear-avoidance, pain-related beliefs, and body-based self-regulation tools (e.g., movement, Graston, percussion massage, and red light therapy).
* Participate in four individual coaching sessions (up to 1 hour each) designed to help them reflect on their experiences, overcome barriers, and integrate the tools into daily life.
* Follow individualized coaching recommendations and provided resources to support each participant's unique engagement with cognitive and body-based tools over the 7-week period, including light journaling, goal setting, and guided reflections.
* Complete brief check-ins every four days to monitor progress, engagement, and self-reported outcomes.

Group and coaching sessions will be recorded and transcribed to support qualitative analysis, allowing researchers to understand how the intervention is experienced and delivered. This will help refine the program for future implementation and scaling. The study prioritizes accessibility, relevance, and peer involvement to address the real-world needs of individuals living with SCI and chronic pain.

DETAILED DESCRIPTION:
Population:

In 2010, it was estimated that over 85,000 Canadians were living with a Spinal Cord Injury (SCI) (Noonan et al., 2012). The severity of the disability associated with SCI varies, depending on the level and completeness of the injury. However, it is common for damage to the spinal cord to result in the loss or severe impairment of mobility, as well as leading to a myriad of secondary health complications (Nash, 2005). Neuropathic pain (NP), experienced by approximately 75% of persons with SCI experience, is one such side effect. Often described as a burning, shooting or stabbing sensation, many who experience it report it being more debilitating than the injury itself (Burke et al., 2017). Currently, treatment options for NP are extremely limited, with pharmaceuticals most often being prescribed to alleviate pain symptoms. Unfortunately, the negative side-effects they elicit are often more unbearable than the actual pain, and with only 30% of individuals reporting a 50% reduction in NP, (Finnerup et al., 2001) many prefer non-pharmaceutical alternatives.(Löfgren & Norrbrink, 2012).

Purpose:

This study aims to evaluate the feasibility and individual-level impact of a 10-week, neuroscience-informed intervention designed to support behavior change in pain self-management among individuals with SCI. The overall study is 10 weeks in duration, with a 7-week intervention and a 3-month post-intervention follow-up data collection.

Hypothesis:

Participants who engage with the program will demonstrate within-person changes in pain-related behaviors, beliefs, and self-regulation strategies. These behavioral shifts are expected to precede reductions in pain interference.

Justification:

Chronic pain after SCI is common and highly disruptive, yet many existing interventions are delivered in group formats that do not flexibly adapt to the diverse and complex needs of individuals. This study addresses that gap by using a personalized, N-of-1 design and a neuroscience-informed approach that supports participants in changing how they think about and respond to pain. Rather than focusing solely on symptom suppression, the program aims to empower participants with tools for self-directed recovery-and to foster the belief that meaningful change, and even healing, is possible.

Objectives:

1. To assess the feasibility, acceptability, and adherence to a 7-week self-management intervention/program focused on pain-related behavior change.
2. To evaluate within-person changes in pain self-management behaviors and beliefs.
3. To examine secondary outcomes, including changes in pain interference, pain severity, and emotional functioning.
4. To understand participants' experiences through qualitative feedback and thematic analysis of open-ended responses.

Research Design and Methods This is a prospective, observational N-of-1 study designed to evaluate the feasibility and individual-level impact of a neuroscience-informed pain self-management intervention for individuals with spinal cord injury (SCI). The study spans 10 weeks, with data collection beginning on Day 1 (20 days prior to the intervention) and continuing every five days throughout the intervention period. A three-month post-intervention follow-up survey is also administered to assess longer-term outcomes.

The intervention itself is seven weeks in duration and is delivered in a non-clinical, coaching-based format. It begins with a 120-minute group education session on Day 22, focused on brain-based pain science and the rationale for behavior change. Participants are then provided with supporting resources to read and view, including the self-help book The Way Out (Gordon, 2022), which introduces principles of Pain Reprocessing Therapy. Additional 120-minute group education sessions are delivered on Day 36 (Optional Body-Based Tools) and Day 64 (Integration, Progress, and Long-Term Self-Management). Up to 60 minutes of peer coaching is offered weekly between group sessions on Days 29-30, 44-45, 50-51, and 57-58. A more detailed explanation of the intervention content and delivery is provided in Section 5.6.

Data are collected via four different online surveys hosted on Qualtrics: Baseline (Day 1), 5-Day Check-In (Days 6, 11, 21, 31, 36, 41, 46, 56, 61, and 66), Mediator Assessments (Days 21, 36, and 51), and Follow-Up (Days 71 and 161). All surveys contain a core set of self-report measures assessing pain interference, pain-related beliefs, emotional functioning, and behavior change processes. The 5-Day Check-In survey includes brief forms of selected measures to reduce participant burden (estimated completion time: 5 minutes), while the other surveys take approximately 20-25 minutes. Open-ended questions are included across all time points to capture qualitative feedback on participant experiences and perceived change.

Statistical Analysis:

Descriptive statistics will be used to assess feasibility and participant characteristics. Within-person change will be evaluated using repeated-measures analyses and time-series plots. Exploratory correlations will examine relationships between engagement and outcome change. Qualitative data will be thematically analyzed to capture participant perspectives, experiences, and perceived mechanisms of change.

ELIGIBILITY:
You can participate in this study if you:

* Have a spinal cord injury (SCI) from a traumatic or non-traumatic cause, experiencing neuropathic/chronic pain
* Are age 18 years or older, and living in Canada
* Can read, speak, and understand English, and have reliable internet access
* Can commit to 10 weeks of data collection (a check-in every 5th day) starting 3 weeks prior to the 7-week intervention, and a 3-month post-intervention follow-up survey.

You cannot participate in this study if you:

* Have an SCI or dysfunction from congenital (e.g., spina bifida), or, other neurological conditions (e.g., MS).
* Are currently participating in CBT or other pain-focused therapy
* Are unwilling or unable to keep pain-related medication stable for the 10-week study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral Change (Engagement / Adherence) | From day 1, every 5 days until the end of the intervention (day 66). Then post intervention (day 71) and 3-month follow-up (day 161).
  Time spent using pain relief tools.
Brief Pain Inventory - Interference | 7-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161). 1-item short form asked on 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66).
  A 7-item self-report measure assessing how pain interferes with daily activities, including general activity, mood, walking ability, work, relationships, sleep, and enjoyment of life.
  A single-item short form will be used for 5-day check-ins.

SECONDARY OUTCOMES:
Brief Pain Inventory - Severity. | 4-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161). 1-item short form asked on 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66).
  A 4-item self-report measure assessing pain intensity at its worst, least, average, and current levels over the past 24 hours, using a 0-10 numeric rating scale. A single-item short-form ("how sever is your pain today") is provided for 5-day check-ins.
Douleur Neuropathique 4 (DN4) | 7-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161). 1-item short form asked on 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66).
  A self-administered screening tool for neuropathic pain, consisting of 7 items assessing sensory descriptors and physical signs. A score of ≥3 suggests neuropathic pain. A single item short-form is provided for 5-day check ins.
  7-item score: Minimum value = 0. Maximum value = 7
  1-item short form: Min. = 0, Max =1.
SOPA-Emotions (Short Form) | 5-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161). 1-item short form asked on 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66).
  A subscale of the Survey of Pain Attitudes assessing beliefs that emotions such as anger and depression influence pain. Higher scores reflect stronger emotional-pain belief endorsement. A single item short-form is provided for 5-day check ins.
  5-item score: Min. = 0, Max = 4 (mean of 5 questions)
  1-item short-form score: Min. = 0, Max =1
Pittsburgh Sleep Quality Index (PSQI) | 19-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161). 1-item short form asked on 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66).
  A 19-item self-report questionnaire assessing sleep quality and disturbances over the past month. It yields a global score (0-21), with higher scores indicating poorer sleep quality. A single item short-form is provided for 5-day check ins.
Pain Catastrophizing Scale (PCS) | 13-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161).
  A 13-item self-report measure assessing catastrophic thinking related to pain. It includes subscales for rumination, magnification, and helplessness. Higher scores indicate greater catastrophizing.
  PCS total score = sum of all 13 items (0-52).
Pain Self-Efficacy Questionnaire (PSEQ) | 10-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161).
  A 10-item self-report measure assessing confidence in performing daily activities despite pain. Higher scores indicate greater pain-related self-efficacy.
  PSEQ score = sum of all 10 items (0-60).
Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS) | 12-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161).
  A 12-item self-report measure assessing satisfaction and frustration of the psychological needs for autonomy, competence, and relatedness. Higher scores reflect greater need satisfaction or frustration.
  Scoring: 1 - 5 (mean of items)
Tampa Scale of Kinesiophobia (TSK-11) | 11-item measure asked: Baseline (day 1), Longer form survey (days 21, 36, 51) and post intervention (days 71, 161).
  An 11-item self-report measure assessing fear of movement or re-injury due to pain. Higher scores indicate greater Kinesiophobia.
  Scoring: Total = sum of all (11-44).
Subjective Happiness Scale (SHS): | 4-item measure asked: Baseline (day 1) and post intervention (days 71, 161). 1-item short form asked: 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66) and longer form survey (days 21, 36, 51).
  A 4-item self-report measure assessing global subjective happiness. Respondents rate their overall happiness and how they compare to peers. Higher scores reflect greater subjective happiness.
  4-item measure scoring: 1 - 7 (mean of 4-items).
  1-item measure: 1-7
UCLA Loneliness Scale (Short Form) | This single-item measure will be asked if every survey: Baseline (day 1), 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, Longer form survey (days 21, 36, 51) and post intervention (days 71, 161).
  A brief self-report measure assessing perceived social isolation and loneliness. Higher scores indicate greater feelings of loneliness. Question 4 (single item).
  Scoring: 1 - 4.
PROMIS Anger (Short Form) | 5-item measure asked: Baseline (day 1) and post intervention (days 71, 161). 1-item short form asked: 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66) and longer form survey (days 21, 36, 51).
  A self-report measure assessing the frequency and intensity of angry feelings over the past 7 days. 5-items. Higher scores indicate greater anger-related distress. A single item short-form is provided for 5-day check ins.
  Scoring: sum of 8-items (8-40) converted to T-score
  - short form 1-item (1-5) converted to T-score
PROMIS Anxiety (Short Form) | 8-item measure asked: Baseline (day 1) and post intervention (days 71, 161). 1-item short form asked: 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66) and longer form survey (days 21, 36, 51).
  A self-report measure assessing symptoms of anxiety, such as fear, worry, and hyperarousal, over the past 7 days. 8-items. Higher scores indicate greater anxiety. A single item short-form is provided for 5-day check ins.
  Scoring: sum of 7-items (7-35) converted to T-score.
  - short form 1-item (1-5) converted to T-score.
PROMIS Depression (Short Form) | 8-item measure asked: Baseline (day 1) and post intervention (days 71, 161). 1-item short form asked: 5-day check-ins (days 6, 11, 16, 26, 31, 41, 46, 56, 61, 66) and longer form survey (days 21, 36, 51).
  A self-report measure assessing depressive symptoms such as sadness, hopelessness, and loss of interest over the past 7 days. 8 items. Higher scores indicate greater depressive symptom severity. A single item short-form is provided for 5-day check ins.
  Scoring: sum of 8-items (8-40) converted to T-score
  - short form 1-item (1-5) converted to T-score
Patient Global Impression of Change (PGIC) | PGIC will be asked post intervention (days 71, 161).
  A single-item self-report measure in which participants rate their overall perception of change in health status since beginning an intervention. Higher scores indicate greater perceived improvement.
  Scoring: 1-7.
Treatment Satisfaction Questionnaire | Treatment Satisfaction Questionnaire will be asked post intervention (days 71, 161).
  A self-report measure assessing participants' satisfaction with various aspects of the intervention, including perceived effectiveness, ease of use, and overall experience. Higher scores indicate greater satisfaction.
  Scoring: 4-items mean score (1-5).
Custom: Confidence in managing pain | This Custom Confidence question will be asked post intervention (days 71, 161).
  Single item open ended question to capture participant's confidence in self-managing their pain following the intervention.
  Scoring: 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Martin Ginis, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared due to concerns regarding participant privacy and confidentiality, particularly given the small and potentially identifiable nature of the spinal cord injury community in Canada. Additionally, the data include sensitive health information that may pose risks if re-identified. The current ethics approval and participant consent do not permit public sharing of individual-level data.